CLINICAL TRIAL: NCT04792983
Title: Cognition and the Immunology of Postoperative Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Deborah Culley, MD, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2019P000577
Record Dates: First submitted 2021-02-26; First posted 2021-03-11 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Impairment; Frail Elderly Syndrome; Delirium; Surgery
Keywords: postoperative health outcomes; older surgical patients; delirium; spine surgery
MeSH Terms: conditions — Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, isolated white blood cells, and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older (≥ 65 years of age): Older surgical patients presenting for elective spine surgery.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study with no interventions.

SUMMARY:
This research will test the hypothesis that immune system disequilibrium / dysfunction explains why preoperative cognitive impairment is a strong predictor of postoperative morbidity in older surgical patients. The investigators propose that cognitive impairment influences surgical morbidity because of underlying immune disequilibrium / dysfunction (risk marker) and that this shapes the immune response to surgery and defines immunological hallmarks of postoperative morbidity (disease marker). The overarching goal of this application therefore is to define and better understand the clinical immunology underlying the relationship between cognition and geriatric surgical morbidity.

DETAILED DESCRIPTION:
This project is designed as a prospective, single-center observational study. The cohort will consist of 600 consenting subjects ≥ 65 years of age that agree to have a study investigator speak with them during their preoperative evaluation prior to elective spine surgery. These ages are chosen as significant clinical data demonstrate increased cognitive impairment in community dwelling elders. Eligibility criteria include: patients ≥ 65 years of age with an American Society of Anesthesiologists (ASA) physical status classification of I-III presenting for elective spinal surgery. Exclusion criteria will include history of stroke (not including transient ischemic attacks, or TIAs) or brain tumor, a history of autoimmune disorders, medications likely to significantly impact inflammation (e.g. steroids), current infection, uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and or inability to speak, read, or understand English.

Patients will be introduced to the study through a flyer provided to them as part of a packet from their surgeon's office. A study team member will speak with those who have agreed during their preoperative evaluation to discuss studies from the department of Anesthesiology and satisfy eligibility criteria. After obtaining informed verbal consent over the telephone, study staff will gain information about the patient's age and years of education. Study staff will conduct the following preoperative measures over the telephone: the Geriatric Depression Scale-Short (GDS), the Beck Anxiety Inventory (BAI), the Visual Analog Scale for Pain (VAS), the Fatigue, Resistance, Ambulation, Illness, and Loss of Weight scale (FRAIL), Instrumental Activities of daily living (IADLs), the Brief Pain Inventory (BPI), the World Health Organization Disability Assessment Schedule (WHODAS). In addition, all patients will be asked if they've had a fall within the last 6 months, whether they've been evaluated for a change in memory or thinking, who accompanied them to their appointment, their employment status and their living situation (alone, institutionalized, living with family members), and whether they have ever tested positive for COVID-19 in a patient survey. The study staff will administer the Montreal Cognitive Assessment (MOCA) simple cognitive screening tool that takes less than 10 minutes to complete and has little or no education, language, or race bias. Frailty will be measured using the Frail Scale. Other measures of cognitive impairment will be obtained by study staff through: documentation on the patient's standard preoperative form, patient or informant report of diagnosis or evaluation for cognitive impairment or memory concerns, and systematic medical record review. Each enrolled patient will be advised to expect a follow up telephone up to 3, 6, and 12- months after surgery to verify data elements and reassess functional outcome.

Delirium will be assessed prospectively once per day on postoperative days 1, 2, and/or 3 by a trained study team member using the Confusion Assessment Method [CAM] if the patient remains in the hospital and agrees to the evaluation. Delirium by chart review and CAM-ICU scores from the nursing staff will also be documented. Delirium is most common on postoperative days 1-3 and the CAM is a well-validated measure of delirium in surgical patients. To evaluate cognition and functional status, the MOCA and the WHODAS will be administered 3, 6, and 12- months postoperatively by study staff over the telephone if the patient can be contacted and continue to agree to participate. The investigators will also collect information on secondary outcomes including whether they had a surgical procedure, time to postoperative anesthesia care unit (PACU) discharge, discharge to place other than home (rehabilitation, skilled nursing facility), hospital length of stay (LOS), 30-day reoperation or readmission rate, and 30-day, 6-month, and 1-year mortality when available. These outcomes are recorded in the medical record, the BWH Balanced Scorecard, an electronic database of all hospitalized patients that tabulates 31 elements of the hospital event, or the Brigham and Women's Hospital BWH Research Patient Database Enhanced Query. Data will also be confirmed by a follow up telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years of age
* American Society of Anesthesiologists (ASA) physical status of I-III
* Scheduled for elective spine surgery.

Exclusion Criteria:

* History of stroke (not including transient ischemic attacks, or TIAs)
* History of brain tumor
* History of autoimmune disorders
* Medications likely to significantly impact inflammation (e.g. steroids)
* Current infection
* Uncorrected vision or hearing impairment
* limited use of the dominant hand (limited ability to draw)
* inability to speak, read, or understand English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The cohort will consist of 600 consenting subjects ≥ 65 years of age who present for preoperative evaluation prior to elective spine surgery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
MOCA Score, Delirium, and Plasma Inflammatory Mediators | 5 years
  The investigators will evaluate correlations between preoperative cognition, as measured by the Montreal Cognitive Assessment (MOCA, minimum score 0 maximum score 30, with higher scores suggesting better cognitive performance) with the development of postoperative delirium and measure preoperative and postoperative plasma inflammatory markers by ELISA to identify whether they correlate with either the MOCA score and/ or the development of postoperative delirium.
MOCA Score, Delirium, and the Cellular Immune Response | 5 years
  The investigators will evaluate correlations between preoperative cognition as measured by the Montreal Cognitive Assessment (MOCA, minimum score 0 maximum score 30, with higher scores suggesting better cognitive performance) with the development of postoperative delirium and measure preoperative and postoperative monocyte immune gene transcriptome ex vivo to identify whether they correlate with either the MOCA score and/ or the development of postoperative delirium.
MOCA Score, Delirium and Extracellular Vesicle Immune Responses to Surgery. | 5 years
  The investigators will evaluate correlations between poor preoperative cognition as measured by the Montreal Cognitive Assessment (MOCA, minimum score 0 maximum score 30, with higher scores suggesting better cognitive performance) with the development of postoperative delirium and measure preoperative and postoperative proteins found in circulating extracellular vesicles by ELISA to identify whether they correlate with either the MOCA score and/ or the development of postoperative delirium.

SECONDARY OUTCOMES:
Newly diagnosed perioperative health complications | Up to 30 days after the surgical procedure
  Newly diagnosed Myocardial Infarction, congestive heart failure (CHF), Cardiac Arrest, Arrythmia, Pneumonia, pulmonary embolism (PE), Reintubation, Stroke, Delirium, Coma>24h, deep wound infection,Superficial wound infection, Sepsis, Renal Failure, urinary tract infection (UTI), Reoperation, deep vein thrombosis (DVT), intensive care unit (ICU) admission following the subjects initial surgical procedure.
Discharge location (Home vs. other than home) on the day of patient discharge from hospital | Up to 30 days after the surgical procedure
  Whether the patient was discharge to their home or discharged to a place other than home such as rehabilitation center or skilled nursing facility.
30 day mortality | 30 days after surgical procedure
  Patient mortality 30 days after surgical procedure
30 day re-operation or readmission | 30 days after surgical procedure
  Patient readmission to the hospital or reoperation 30 days after surgical procedure
6 month mortality | 6 months after surgical procedure
  Patient mortality 6 months after surgical procedure
1 year mortality | 1 year after surgical procedure
  Patient mortality 1 year after surgical procedure
Cognitive health outcome | 3, 6, and 12-months after surgical procedure.
  Montreal Cognitive Assessment (MOCA, minimum score 0 maximum score 30, with higher scores suggesting better cognitive performance) measured approximately 3, 6, and 12-months following the patient's surgical procedure if the participant is willing to participate.
Functional health outcome | Between 6 and 12-months after surgical procedure.
  Functional health outcome measured with the World Health Organization Disability Assessment Score (WHODAS, 12-item, minimum score 0 maximum score 110 with higher score reflecting more disability) approximately 6 months to 1 year following the patient's surgical procedure if the participant can be contacted by followup phone call and is willing to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Crosby, MD, Principal Investigator — Brigham & Women's Hospital; Harvard Medical School
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided